CLINICAL TRIAL: NCT03503487
Title: Surgical Planning and Informed Consent
Acronym: SPLICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Principal Investigator, Eleonora Orena, Psychologist, Neuroscientist researcher, Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SPLICE
Record Dates: First submitted 2018-04-04; First posted 2018-04-19 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Communication; Feedback, Psychological; Health Knowledge, Attitudes, Practice; Humans; Informed Consent; Neurosurgery; Patient Compliance; Patient-Centered Care; Physician-Patient Relations; User-Computer Interface
MeSH Terms: conditions — Communication; Behavior; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Patients receiving standard informed consent procedure before intervention
- Planner 1 (Experimental): Patients receiving 3D informed consent procedure before intervention with Surgical Theater
  Interventions: Other: 3D informed consent
- Planner 2 (Experimental): Patients receiving 3D informed consent procedure before intervention with Vesalius
  Interventions: Other: 3D informed consent

INTERVENTIONS:
Other: 3D informed consent — Patients were given an informed consent with the aid of a 3D immersive surgical planner (either a Surgical Theater or Vesalius)
  Arms: Planner 1; Planner 2

SUMMARY:
New devices for anatomic studies and 3-D visualization have proven to be useful for pre-operative surgical planning and intra-operative procedures; the hypothesis of our study is that, in this specific case scenario, Surgical Theater and Vesalius (two devices available at the Besta NeuroSim Center, Foundation I.R.C.C.S. Neurological Institute Carlo Besta) can improve doctor-patient communication during the process of obtaining informed consent: through tridimensional representation of anatomic structures of the brain, these devices are able to help patients understand better their own anatomy and the surgical approach to their disease.

The aim of our study is therefore to understand whether this high-technology 3D planning, used as a tool to optimize patient-doctor communication, can effectively improve patients' understanding of the disease and the surgical procedure they will be going through (for which they are supposed to sign the consent), as well as the benefits, the risks and all the possible complications that can derive form surgery.

Surgical Theater and Vesalius may be of great help: thanks to the case-specific 3D reconstruction of the patient's anatomy, the explanation of the surgical procedure could be customized for each different person, considering that anyone has certain unique individual features that a regular standardized system could not possibly take into account.

DETAILED DESCRIPTION:
Informed consent is the authorisation of an activity based on the understanding of what that activity entails in the absence of control by others. In surgery this process needs the comprehension of the benefits and the risks of the operation. Despite this, it has been argued that most surgeons do not devote adequate importance and time to this step in their daily practice; sometimes they are just afraid of scaring the patients with too many unnecessary details. Surgeons then might hide themselves behind legal booklets that should provide all information; too often though, patients do not fully realise their diseases and the possible outcomes.

New devices for anatomical studies and 3D visualization have proven to be useful for preoperative surgical planning and intra-operative procedures; the hypothesis of our study is that Surgical Theater and Vesalius (two new-generation, immersive, 3D imaging visualizers) can improve doctor-patient communication during the process of obtaining informed consent: through the tridimensional representation of anatomic structures of the brain, these devices are able to help patients better understand their anatomy, the surgical approach for their disease and possible complications.

In a prospective, randomized controlled pilot study, 40 patients undergoing neurosurgery for intracranial tumours were enrolled. Patients' cognitive function, verbal comprehension and memory were assessed before being enrolled. All groups initially underwent the standard informed consent process. Then the experimental groups received a second informed consent process with the aid of surgical planners, while the control group went through to a second round of standard informed consent. Questionnaires about appreciation, anxiety, and perceived and objective comprehension (on pathology, surgery, complications) were given.

Tridimensional surgical planners may be of great help in improving how technical information is conveyed to patients when consented for surgery. Considering that every individual has unique features, a standardised method cannot be taken into account, therefore, thanks to the case-specific 3D reconstruction of the patient's anatomy, the explanation of the surgical procedure can be customized for every patient. Using new 3D technologies is expected to reduce patients' anxiety and to improve the understanding of their conditions and the possible consequences related to any treatment options.

ELIGIBILITY:
Inclusion Criteria:

* having a cerebral tumor
* no visual/auditory deficit
* no psychiatric illness
* italian mother-tongue

Exclusion Criteria:

* younger than 18 or older than 70
* pre-existing perceptual deficit and/or psychiatric illness
* not italian mother-tongue

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the comprehension of the benefits/risks of the intervention | 1 year
  Comprehension of the benefits/risks of the intervention evaluated through a ad hoc questionnaire

SECONDARY OUTCOMES:
Level of patient's anxiety | 1 year
  Anxiety score pre- and post- informed consent as assessed with the State-Trait Anxiety Inventory (STAI) Y-1 and Y-2

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Perin, MD, PhD, Principal Investigator — Foundation IRCCS Neurologic Institute Carlo Besta
Locations (1):
- Foundation IRCCS Neurologic Institute Carlo Besta, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perin A, Galbiati TF, Ayadi R, Gambatesa E, Orena EF, Riker NI, Silberberg H, Sgubin D, Meling TR, DiMeco F. Informed consent through 3D virtual reality: a randomized clinical trial. Acta Neurochir (Wien). 2021 Feb;163(2):301-308. doi: 10.1007/s00701-020-04303-y. Epub 2020 Apr 3. PMID 32242272